CLINICAL TRIAL: NCT04345133
Title: Effect of Undersized Drilling Upon the Primary and Secondary Stability of Immediate Conical Implants in the Esthetic Maxillary Sector
Brief Title: Effect of Undersized Drilling Upon the Immediate Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Carabobo (Other)
Responsible Party: Principal Investigator, Alejandro Sierra-Rebolledo, Associate Professor, University of Carabobo
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UCarabobo
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Implant Stability
Keywords: Primary Stability; Secondary Stability; Undersized Drilling

STUDY DESIGN:
Intervention Model Description: Comparative
Who Masked: Participant
Masking Description: No informaron about sequence of drilling was used to insert the implants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Undersized Drilling Group (Active Comparator): Exposed patients to the reduction of the final drill dimensions at the insertion implants protocol sequence
  Interventions: Device: Dental Implants Insertion Drilling Sequence
- Conventional Drilling Group (Other): Group with the conventional protocol recommended by the manufacturer
  Interventions: Device: Dental Implants Insertion Drilling Sequence

INTERVENTIONS:
Device: Dental Implants Insertion Drilling Sequence — Drilling sequence protocol to insert immediate Dental Implants at the Maxilla.

SUMMARY:
OBJECTIVE:

evaluate the effect of undersized drilling upon the primary and secondary stability of immediate implants placed in the anterior sector maxilla.

PATIENTS AND METHODS Study design A randomized comparative clinical trial was carried out. Thirty conical MIS C1 grade 23 titanium alloy (Ti 6Al 4V Eli) implants with a rough surface subjected to dual acid etching and sandblasting, measuring 3.75 mm in maximum diameter and 13 mm in length (MIS® Implants Technologies, Ltd. Bar Levi, Israel), were placed immediately after removal a anterior maxillary tooth in a series of patients treated in the clinic of the Master of Dentistry and Dental Implantology (Santa María University, Dental School, Caracas, Venezuela). The study was approved by the local Ethics Committee.

Patient selection To enrolled in the study, patients had to comply the inclusion/exclusion criteria established to the study: over 18 years of age with indication of one or more immediate implants in the anterior maxilla; no history of ischemic heart disease, uncontrolled diabetes, coagulation disorders, head or neck radiotherapy, intravenous bisphosphonates or uncontrolled periodontal disease. Based on a CTCB evaluation, the teeth involved should have presence of bone ≥ 5 mm from the tooth apex to the lower cortical layer of the nasal fossa / maxillary sinus and no vertical defects greater than 4 mm at the buccal or palatine alveolar crest. Also, patients must have capacity to understand the study protocol and fill consent form to participation in the study.

Study procedure Two operators calibrated for immediate implant placement performed minimally traumatic tooth extraction following local infiltrating anesthesia with 4% articaine and 1:100,000 epinephrine (Artheek® 4%, New Stetic S.A.; Antioquia, Colombia). After evaluating the integrity of the bone walls, drilling sequence was established on a randomized basis.

Conventional drilling (CD) sequence:

* Marking drill ∅1.9 mm at 1500 rpm
* Pilot drill ∅ 2.4 mm and 13 mm in length at 800 rpm.
* Twist drill ∅3 mm at 400 rpm.

Undersized drilling (UD) sequence:

Marking drill ∅1.9 mm at 1500 rpm Pilot drill ∅ 2.4 mm and 13 mm in length at 400 rpm. Implant insertion A surgical motor (MCU MIS, model M0132, W&H, Burmoos, Austria) with a 20:1 reducing implant handpiece was used to insert the implants at 20 rpm and applying a torque of 10 Ncm. Following placement of the implant in the bed, manual insertion was continued to reach the final implant position, established as 4 mm from the gingival margin.

Study variables Two torque meters (MIS® Implants LTD, models MT-RI040 and MT-RT070, Bar Levi, Israel) were used to insert and sequentially measure the maximum IT reached on positioning the implant in the socket. A Smart-peg Nro 49 model 100480 was fitted to the connection of each implant and an Osstell ISQ® (SN 4669 Osstell AB, Goteborg, Sweden) was used to perform RFA analysis and obtain corresponding ISQ value at insertion time (RFA1). A 4 mm height healing screw was used to seal the implant, and then additional RFA measurements was made at 6 week (RFA2) and 12 week (RFA3) post-implantation

ELIGIBILITY:
Inclusion Criteria:

indication of one or more immediate implants in the anterior maxilla; No history of ischemic heart disease, No History of uncontrolled diabetes, No coagulation disorders, No head or neck radiotherapy

Exclusion Criteria:

Periodontal Disease. History of EV or Oral Bisphosphonate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-12-17 (Actual); Study Completion 2018-03-17 (Actual)

PRIMARY OUTCOMES:
Insertion Torque | at baseline, through study completion in average 1 year
  Maximum torque in N.cm obtained during insertion of the implant
RFA Implant Stability | at baseline, through study completion in average 1 year
  Implant Stability measure by Radio-Frequency Analysis.

SECONDARY OUTCOMES:
RFA2 Implant Stability | 6 weeks after baseline, trough study completion in average 1 year
  Implant Stability measure by Radio-Frequency Analysis 6 weeks later
RFA3 Implant Stability | 12 weeks after baseline, trough study completion in average 1 year
  Implant Stability measure by Radio-Frequency Analysis 12 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Sierra-Rebolledo, DDS, Principal Investigator — University of Carabobo, Faculty of Dentistry

IPD SHARING:
Plan to Share IPD: No
The study protocol is included in the medical records of the postgraduate degree and there are identity protection policies.

REFERENCES:
- [Background] Sierra-Rebolledo A, Allais-Leon M, Maurette-O'Brien P, Gay-Escoda C. Primary Apical Stability of Tapered Implants Through Reduction of Final Drilling Dimensions in Different Bone Density Models: A Biomechanical Study. Implant Dent. 2016 Dec;25(6):775-782. doi: 10.1097/ID.0000000000000479. PMID 27540846